CLINICAL TRIAL: NCT06162052
Title: Impact of a Telerehabilitation Program With Technology Enhancement on Post-burn Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-0331
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Standard of Care group (SOC) (Experimental): Participants will receive standard of care education by the physical or occupational therapist regarding performance of the prescribed movements prior to discharge. Participants will complete the study about 6 months after discharge.
  Interventions: Other: Tele-Rehabilitation
- A Standard of Care group (SOC) combined with technology enhancement (Experimental): Participants will receive standard of care education by the physical or occupational therapist regarding performance of the prescribed movements prior to discharge. Participants will undergo additional training in the use of a goniometer to measure range of motion at home and record the measurement once a week for 6 months. Participants will engage in 4 virtual sessions as well as wear a Fitbit
  Interventions: Other: Tele-Rehabilitation

INTERVENTIONS:
Other: Tele-Rehabilitation — Technology will be used to enhance rehabilitation.

SUMMARY:
The purpose of this study is to examine the effect of participating in a tele-rehabilitation program after a burn.

DETAILED DESCRIPTION:
This is a prospective single center randomized trial comparing a traditional approach to physical therapy to a technology-enhanced approach following a burn. We hypothesize that with the implementation of a novel telerehabilitation program incorporating technology enhancement, range of motion and quality of life can be improved. To test the hypothesis in future grant applications, this pilot study will be used to determine feasibility, collect preliminary data, vet endpoints, and gain patient feedback. To achieve these necessary goals, we will compare two methods of supporting home performance of prescribed physical and occupational therapy: Standard (S): patients will be equipped with paper instructions for their physical therapy exercises; and Technology-Enhanced (TE) support: patients will be given paper instructions, set up with a habit and productivity application (Avocation) that gamifies tasks and tracks achievements, a Fitbit activity tracker, a logbook, and have virtual movement therapy once weekly with an exercise physiologist for a total of four weeks.

Specific Aim 1: To determine whether range of motion is altered with TE. Range of motion in the affected joint(s) will be measured by goniometry (self-reported by patient and measured by study staff in the clinic)

Specific Aim 2: To determine whether TE with prescribed movement affects scar, pain, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults: ≥18 to ≤79 years of age
* Not participating in another interventional trial
* Admitted to the Blocker Burn Unit for treatment of initial burn
* Subject is able and willing to follow the protocol requirements
* Burn wound / scar / contracture occurring across at least one joint.
* Has regular access to smart phone, tablet, or computer with internet access.

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigator or physician, would place the subject at increased risk for participation.
* Concurrent participation on another interventional clinical trial
* History of prior non-compliance or the presence or history of psychiatric condition (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.
* Patients without internet access.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in range of motion, measured with a goniometer | Prior to planned discharge or during first week post- discharge (Baseline), and at clinic visits approximately 1, 3, & 6 months after discharge (±15 days, each timepoint)
  Patient will be asked to bend the affected joint, and the goniometer held next to the joint to measure the angle. The range of motion for the opposite joint will be measured as well.

SECONDARY OUTCOMES:
Scar Volume | Prior to planned discharge or during first week post- discharge (Baseline), and at clinic visits approximately 1, 3, & 6 months after discharge (±15 days, each timepoint)
  3D photo taken with LifeViz 3DII camera.
Elasticity, color, temperature, trans epidermal water loss, and scar thickness | Prior to planned discharge or during first week post- discharge (Baseline), and at clinic visits approximately 1, 3, & 6 months after discharge (±15 days, each timepoint)
  Measured with Dermalab combo (Cortex Technology, Denmark); each probe is held with constant pressure on the skin or scar surface for one minute; multiple measures are conducted to reduce variability.
Blood Flow | Prior to planned discharge or during first week post- discharge (Baseline), and at clinic visits approximately 1, 3, & 6 months after discharge (±15 days, each timepoint)
  A laser speckle device will be used to measure blood flow without contact.
Patient and Observer Scar Assessment Scale v2.0 | Prior to planned discharge or during first week post- discharge (Baseline), and at clinic visits approximately 1, 3, & 6 months after discharge (±15 days, each timepoint)
  The scale consists of six items rated from 1 to 10, where 1 is "normal skin" and 10 is the "worst imaginable scar". The observer (i.e., investigator) evaluates scar vascularity, pigmentation, thickness, relief, pliability, and surface area. The scores of each of the six items are summed for a total score (range 6 to 60).
Pain Visual Analog Scale (VAS) Score | Prior to planned discharge or during first week post- discharge (Baseline), and at clinic visits approximately 1, 3, & 6 months after discharge (±15 days, each timepoint)
  Pain severity scores at rest will be assessed by use of a visual analog scale (VAS; 0 = no pain, 100 = worst pain imaginable).
Post Interview | 6 months (± 2 weeks) post discharge
  At the conclusion of each patient's participation, they will meet with an investigator or delegated study staff for a brief non-structured interview to discuss participation in the study including improvements for follow-up studies.
Overall Activity | Months 2, 4, and 5 (+15 days, each timepoint) in addition to 1, 3, & 6 months after discharge.
  To be captured via Fitbit on a daily basis to gauge overall activity. These data will be correlated with the pain scale as reduced activity is associated with pain.
Itch Scale | Prior to planned discharge or during first week post- discharge (Baseline), and at clinic visits approximately 1, 3, & 6 months after discharge (±15 days, each timepoint)
  A Visual Analog Scale will be used for patients to rate their itch from 0 to 100. (VAS; 0 = no itch, 100 = worst itch imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Finnerty, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No